CLINICAL TRIAL: NCT05175339
Title: Long-term Impact in Intensive Care Survivors of Coronavirus Disease-19
Brief Title: Long-term Impact in Intensive Care Survivors of Coronavirus Disease (COVID-19)
Acronym: AFTERCOR
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00276578
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Investigator seeks to evaluate the long term neurological and pulmonary sequelae of COVID-19.

DETAILED DESCRIPTION:
Recent data suggests that survivors of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or (COVID-19) report adverse health status, including neurological and cognitive deficits and impaired pulmonary function, even months after discharge. Adult COVID-19 survivors after ICU stay, who are noted to have increased mortality and organ failure, are at higher risk of long-term disabilities and impaired quality of life. This study is one branch of a multi-site study coordinated by Gilead Sciences, in which participants who were critically ill with COVID-19 will be followed at three and nine months after discharge to test pulmonary function, cognitive function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected or laboratory confirmed COVID-19 infection by real-time PCR
* Admission to an intensive care unit for COVID-19 and discharge

Exclusion Criteria:

* Pregnancy
* Participants unable to complete long-term follow-up due to logistical problems
* Participant paralyzed before being admitted to hospital for COVID-19
* History of pulmonary resection
* Previous pulmonary transplant
* Documented advanced neurologic order for which the patient is unable to carry out 6 minute walk test
* Documented psychiatric disease for which the patient is unable to carry out interview

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study population includes polymerase chain reaction (PCR) confirmed COVID-19 patients at Johns Hopkins Hospital and UT Houston Health Science Center who required intensive care unit admission for COVID-19 management.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary quality of life as assessed by St. George's Respiratory Questionnaire | 3 months and 9 months post-discharge
  St. George's Respiratory Questionnaire measures quality of life associated with chronic respiratory diseases. It has been used in various reports of long-term impact of acute respiratory distress syndrome. Scores for each domain range from 0 to 100, with a lower score indicating better pulmonary-specific quality of life.
Change in pulmonary capacity as assessed with forced vital capacity | 3 months and 9 months post-discharge
  Forced vital capacity will be measured with pulmonary function testing.
Change in pulmonary capacity as assessed with forced expiratory volume | 3 months and 9 months post-discharge
  Forced expiratory volume will be measured with pulmonary function testing.
Change in pulmonary capacity as assessed with forced expiratory ratio | 3 months and 9 months post-discharge
  Forced expiratory ratio will be measured with pulmonary function testing.
Change in cardiopulmonary and musculoskeletal strength as assessed by a six minute walk test | 3 months and 9 months post-discharge
  Six Minute Walk Test provides an objective measure of cardiopulmonary and musculoskeletal function by recording distance (in meters) walked in six minutes.
Evaluation of residual pulmonary pathology as assessed by a chest x-ray | 3 months post-discharge
  Chest X-Ray will be used in the evaluation of residual pulmonary pathology.
Evaluation of residual pulmonary pathology as assessed by a chest x-ray | 9 months post-discharge
  Chest X-Ray will be used in the evaluation of residual pulmonary pathology.

SECONDARY OUTCOMES:
Change in cognitive function as assessed by the Montreal Cognitive Assessment (MoCA) | 3 months and 9 months post-discharge
  Montreal Cognitive Assessment assesses cognitive impairment and recovery by evaluating attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
Change in cognitive function as assessed by BrainCheck | 3 months and 9 months post-discharge
  BrainCheck is a computer-based test that assesses a variety of cognitive domains. For each individual test, the BrainCheck platform provides standard scores and percentile ranks. Additionally, the platform provides a composite score for an overall assessment of cognitive function. These scores are adjusted for age, derived from a normative database ranging from ages 10 to 99. Patient scores that fall within a range of one standard deviation above and below the mean indicate "normal" cognitive function. Low scores outside of this range suggest cognitive impairment.
Change in depressive symptoms as determined by PHQ-9 | 3 months and 9 months post-discharge
  PHQ-9 is a nine question screening tool that aids in the diagnosis and symptom tracking of depression. The possible range of scores is 0-27. Scores from 0-4 represent minimal depression, 5-9 represents mild depression, 10-14 represents moderate depression, 15-19 represents moderately severe depression, and 20-27 represents severe depression.
Change in prevalence of anxiety symptoms as determined by GAD7 | 3 months and 9 months post-discharge
  GAD7 is a seven question tool used to measure severity of generalized anxiety disorder. Responses are measured on a scale from 0-21, with higher scores representing more severe anxiety.
Change in quality of life as assessed by Fatigue Severity Scale | 3 months and 9 months post-discharge
  Fatigue severity scale measures the severity of fatigue and its impact on a person's lifestyle using a 9-item scale. Each item is scored on a 7 point scale. Total scores range from 9-63 with higher scores representing greater fatigue severity.
Change in quality of life as assessed by Pain, Enjoyment of life, and General activity (PEG) screening tool | 3 months and 9 months post-discharge
  PEG tracks severity of pain and impact on quality of life using three questions. The mean response is calculated from the three items. Total score ranges from 0-10 with lower scores representing less pain and more favorable quality of life.
Change in post-traumatic stress disorder (PTSD) symptoms with PTSD-5 | 3 months and 9 months post-discharge
  PTSD-5 is a five-question screening tool for identification of post-traumatic stress disorder. Total score ranges from 0-5, with scores of 3 or greater representing probable PTSD.
Neurological assessment with brain MRI | 3 months post-discharge
  Brain MRI to assess clinical and/or subclinical brain injury such as infarcts, hemorrhages, and microhemorrhages.
Change in health-related Quality of Life as assessed by the short form (SF)-36 survey | 3 months and 9 months post-discharge
  The SF-36 survey is a questionnaire that assesses the eight domains of physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, physical energy, and general health perceptions. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Jannelle Molina, Study Director — Gilead Sciences
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Texas Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other institutions. Deidentified information will be shared between the two site locations and with investigators involved in the AFTERCOR trial with Gilead sciences.